CLINICAL TRIAL: NCT03891004
Title: Skin Closure With Tissue Adhesives vs. Subcuticular Suture After Robotic Urogynecologic Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. John Hospital & Medical Center (Other)
Responsible Party: Principal Investigator, Sunetris Fluellen, Principal Investigator, St. John Hospital & Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: StJohnHMedCtr
Record Dates: First submitted 2018-03-18; First posted 2019-03-26 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Surgical Wound; Tissue Adhesion
MeSH Terms: conditions — Surgical Wound; Tissue Adhesions | interventions — Tissue Adhesives

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial comparing skin closure after robotic urogynecologic surgery with tissue adhesive versus subcuticular suture.
Who Masked: Participant, Outcomes Assessor
Masking Description: The evaluators of cosmesis will be blind to the group assignment. The person who will evaluate the scars will be a nurse or medical assistant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Tissue Adhesives Only (Experimental): For the tissue adhesive, we will use Dermabond, which was FDA approved for skin closure in 1998. We will record the length of time of each closure method for comparison, and have patients follow-up at two, six and 12 weeks. At the 12 week visit we will score the appearance of the incision.
  Interventions: Device: Tissue Adhesives
- Subcuticular Suture Closure Method Only (Active Comparator): For the suture arm we will only close the subcuticular layer. We will record the length of time of each closure method for comparison, and have patients follow-up at two, six and 12 weeks. At the 12 week visit we will score the appearance of the incision.
  Interventions: Procedure: Subcuticular Skin Closure

INTERVENTIONS:
Procedure: Subcuticular Skin Closure — We will only close the subcuticular layer with suture
  Arms: Subcuticular Suture Closure Method Only
Device: Tissue Adhesives — No subcuticular closure will be done. Only tissue adhesives applied to the approximated skin
  Arms: Tissue Adhesives Only

SUMMARY:
To compare skin closure via subcuticular suture versus tissue adhesive (Dermabond) in urogynecological robotic surgeries. The primary outcome is incision cosmesis at the 12 week follow up visit. Secondary outcome is the operative time between the two methods of closure.

DETAILED DESCRIPTION:
The purpose of this study is compare skin closure via suture versus tissue adhesive (Dermabond) in urogynecological robotic surgeries. The primary outcome is incision cosmesis. Therefore, if the tissue adhesive is cosmetically comparable to that of sutures, that will be reason to use tissue adhesives over traditional sutures. In these surgeries, there are five to six port sites (compared to fewer for usual laparoscopic procedures) and the procedures are lengthy procedures (average duration about 300 minutes as per recent AUGS/ACOG committee opinion), so if the investigators can show significant time reduction for closure, that should reduce operative time and costs. To the investigators' knowledge, this will be the first study of its kind to make this comparison for urogynecologic robotic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Women, ages 18 years and older, undergoing any urogynecologic robotic procedure at St. John Hospital and Medical Center from March 19, 2018 - November 30, 2018.

Exclusion Criteria:

* We will exclude women with active skin infections as they may contribute to poor wound healing and infections. We will also exclude procedures that are converted to laparotomy.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females as this pertains to skin closure of robotic urogynecology procedures
Enrollment: 47 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Incision Cosmesis | 12 weeks
  Our primary outcome measure is to compare incision cosmesis between the two closure methods at the 12 week postoperative visit. The Stony Brook Scar Evaluation scale is used. A point is awarded in each of the following categories: width, height, color, hatch/suture marks, overall appearance. Poorer cosmesis is indicated by a lower score. Highest score possible is 5 points.

SECONDARY OUTCOMES:
Incision closure time | 30 minutes
  The time of each closure method will be recorded and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- St. John Hospital & Medical Center, Detroit, Michigan, United States